CLINICAL TRIAL: NCT01836653
Title: Randomized Phase II Study of mFOLFOX6 + Bevacizumab or mFOLFOX6 + Cetuximab in Liver Only Metastasis From KRAS Wild Type Colorectal Cancer
Brief Title: Achievement of Improved Survival by Molecular Targeted Chemotherapy and Liver Resection for Not Optimally Resectable Colorectal Liver Metastases
Acronym: ATOM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EPS Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATOM; UMIN000010209 (Other: UMIN)
Record Dates: First submitted 2013-04-14; First posted 2013-04-22 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Liver Only Metastasis From KRAS Exon 2 Wild Type (Under Protocol 1.0-1.2 Edition) and RAS Wild Type (Under Protocol 2.0 Edition) Colorectal Cancer
Keywords: Bevacizumab; Cetuximab; KRAS wild type colorectal cancer; RAS wild type colorectal cancer; liver metastasis
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Cetuximab; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mFOLFOX + Bmab (Experimental): mFOLFOX plus bevacizumab
  Interventions: Drug: Bevacizumab; Drug: L-OHP; Drug: l-LV; Drug: 5-FU
- mFOLFOX + Cmab (Active Comparator): mFOLFOX plus cetuximab
  Interventions: Drug: Cetuximab; Drug: L-OHP; Drug: l-LV; Drug: 5-FU

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/kg intravenously administered over 90 minutes (can be reduced to 30 minutes at the minimum) on day 1 of a 2-week cycle. Liver resection if resectable after 8 cycles or continue until progression of disease.
  Other Names: Avastin
  Arms: mFOLFOX + Bmab
Drug: Cetuximab — 250 mg/m2 intravenously administered over 60 minutes (400 mg/m2 over 120 minutes as the initial dose) on day 1 and day 8 of a 2-week cycle. Liver resection if resectable after 8 cycles or continue until progression of disease.
  Other Names: Erbitux
  Arms: mFOLFOX + Cmab
Drug: L-OHP — 85 mg/m2 intravenously administered over 120 minutes on day 1 of a 2-week cycle. Liver resection if resectable after 8 cycles or continue until progression of disease.
  Other Names: Oxaliplatin
Drug: l-LV — 200 mg/m2 intravenously administered over 120 minutes on day 1 of a 2-week cycle. Liver resection if resectable after 8 cycles or continue until progression of disease.
  Other Names: Levofolinate
Drug: 5-FU — 400 mg/m2 intravenous bolus on day 1 of a 2-week cycle. Liver resection if resectable after 8 cycles or continue until progression of disease.
  Other Names: Fluorouracil
Drug: 5-FU — 2400 mg/m2 continuous infusion over 46 hours on day 1 and 2 of a 2-week cycle. Liver resection if resectable after 8 cycles or continue until progression of disease.
  Other Names: Fluorouracil

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of mFOLFOX6+bevacizumab and mFOLFOX6+cetuximab for liver only metastasis from KRAS Exon 2 wild type (under protocol 1.0-1.2 edition) and RAS wild type (under protocol 2.0 edition) colorectal cancer.

DETAILED DESCRIPTION:
Description: The purpose of this study is to evaluate efficacy and safety of mFOLFOX6+bevacizumab and mFOLFOX6+cetuximab for liver only metastasis from KRAS Exon 2 wild type (under protocol 1.0-1.2 edition) and RAS wild type (under protocol 2.0 edition) colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed colorectal cancer (adenocarcinoma) excluding vermiform appendix cancer and proctos cancer.
2. RAS wild type
3. Synchronous* or metachronous liver limited meitastasis with no extrahepatic desiease

   * shychronous liver limited metastasis with primary lesion less than two thirds of the circumference
   * patients with primary lesion more than two thirds of the circumference can be enrolled after primary resection
4. Patients who has one or more lesion(s) of diameter 1 cm or larger (RECEST v1.1) be able to assess continuously on the basis of the protocol by contrast enhanced CT or contrast enhanced MRI of the liver:

(1)Liver metastases 5 or more (2)Liver metastases with 5 cm or larger in greatest dimension (3)Unresectable considering remaining hepatic function (4)Invasion into all hepatic veins or inferior vena cava (5)Invasion into both right and left hepatic arteries or portal veins 5.No prior chemotherapy for colorectal cancer including hepatic arterial infusion. Excluding postoperative and preoperative chemoradiotherapy except for rectal cancer with synchronous liver metastases. Patients received postoperative chemotherapy containing oxaliplatin have to be enrolled after 24 weeks from the last oxaliplatin administration.

6.No previous treatment including ablation therapy, cryotherapy and chemotherapy for metastases 7.Age at enrollment is >=20 and =<80 years 8.The Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 9.Life expectancy from the day of enrollment is 3 months or longer 10.Major organ functions less than 14 days prior to entry meet the following criteria.

1. Neu >= 1500/mm3
2. Pt >= 10.0x10^4/mm3
3. Hb >= 9.0 g/dL
4. T-bil =< 2.0 mg/dL
5. AST and ALT =< 200 IU/L
6. sCr =< 1.20 mg/dL
7. INR < 1.5
8. Proteinuria =< 2+ 11.Written informed consent

Exclusion Criteria:

1. Previously experienced severe allergic reaction to drugs
2. Receiving anti-platelet drugs (aspirin >= 325 mg/day) or NSAIDs
3. Receiving chronic systemic corticosteroid treatment
4. Surgery/ biopsy with skin incision or traumatic injury with suture less than 14 days prior to entry. Excluding, suture for implanted venous reservoirs with catherter is allowed.
5. Severe postoperative complications (e.g. postoperative infection, anastomic dehiscence or paralytic ileus)
6. Diagnosed as hereditary colorectal cancer
7. Active other malignancies
8. Cerebrovascular disease or symptoms less than 1 year prior to entry
9. Pleural effusion, ascites or cardiac effusion requiring drainage
10. Hemorrhage/bleeding, paralytic ileus, obstruction or ulceration of gastrointestinal tract
11. Perforation of gastrointestinal tract less than 1 year prior to entry
12. Presence of active infection
13. HBs antigen or HCV antibody positive
14. Uncontrolled comorbidity including hypertension, diabetes, arrhythmia, or other diseases (such as cardiac disorder, interstitial pneumonia or renal disorder)
15. Presence of >= grade 2 diarrhea
16. Presence of >= grade 1 peripheral neuropathy
17. Pregnant or lactating women. Women and men with childbearing potential unwilling to use effective means of contraception
18. Psychosis or psychiatric symptoms who are not able to comply with the protocol
19. Any other medical conditions disable to comply with the protocol

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | assessed every 8 weeks, up to 4 years
  assessed by Independent Review Committee

SECONDARY OUTCOMES:
Response rate | assessed every 8 weeks, up to 4 years

OTHER OUTCOMES:
Tumor shrinkage rate at 8 week | assessed at 8 week, up to 8 weeks
Liver resection rate | assessed every 8 weeks, up to 4 years
R0 liver resection rate | assessed every 8 weeks, up to 4 years
  pathologically confirmed R0 liver resection rate
Progression-free survival | assessed every 8 weeks, up to 4 years
  assessed by investigators
Time to treatment-failure | assessed every 2 weeks, up to 4 years
Overall survival | assessed every 2 weeks, up to 4 years
Quality of life | assessed every 16 weeks, up to 1 year
Incidence of adverse events | assessed every 2 weeks, up to 4 years
Progression-free survival among the RAS wild type subpopulation | assessed every 8 weeks, up to 4 years
  All the assessment is repeated for a maximum of 4 years.

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihiko Maehara, MD,PhD,FACS, Principal Investigator — Graduate School of Medical Science, Kyushu University, Department of Surgery and Science; Naohiro Tomita, MD, PhD, Principal Investigator — Hyogo College of Medicine, Department of Surgery; Ichinosuke Hyodo, MD, PhD, Principal Investigator — Tsukuba University, Graduate School of Medicine; Michiaki Unno, MD, PhD, Principal Investigator — Tohoku University, Division of Gastroenterological Surgery
Locations (1):
- EPS Corporation, Shinjuku-ku, Tokyo, Japan

REFERENCES:
- [Derived] Oki E, Emi Y, Yamanaka T, Uetake H, Muro K, Takahashi T, Nagasaka T, Hatano E, Ojima H, Manaka D, Kusumoto T, Katayose Y, Fujiwara T, Yoshida K, Unno M, Hyodo I, Tomita N, Sugihara K, Maehara Y. Randomised phase II trial of mFOLFOX6 plus bevacizumab versus mFOLFOX6 plus cetuximab as first-line treatment for colorectal liver metastasis (ATOM trial). Br J Cancer. 2019 Jul;121(3):222-229. doi: 10.1038/s41416-019-0518-2. Epub 2019 Jul 9. PMID 31285591